CLINICAL TRIAL: NCT07282756
Title: Assessment of Changes in Clinical and Radiological Parameters in Gingival Pockets After Subgingival Application of 1.2% Lovastatin Gel in Combination With SRP Procedure Compared to SRP and Placebo Gel Application in the Treatment of Periodontal Disease in Generally Healthy Non-smokers and Smokers From Central Europe: a Split-mouth Randomized Controlled Trial.
Brief Title: EVALUATION OF THE EFFECTIVNESS OF SUBGINGIVAL APPLICATION OF 1.2% LOVASTATIN GEL AS AN ADJUNCT TO NON-SURGICAL TREATMENT OF PERIODONTITIS IN GENERALLY HEALTHY SMOKERS AND NON-SMOKERS PATIENTS FROM CENTAL EUROPE- A SPLIT-MOUTH RANDOMIZED CONTROLLED TRIAL.
Acronym: RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Silesia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025/6/5/4
Record Dates: First submitted 2025-11-18; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-11

CONDITIONS: Periodontal Diseases; Periodontitis; Periodontal Disease; Smokers
Keywords: periodontitis; statins; lovastatin; smoking; periodontal disease
MeSH Terms: conditions — Periodontal Diseases; Periodontitis; Smoking | interventions — Lovastatin

STUDY DESIGN:
Intervention Model Description: After the SRP procedure is applied within the qualified gingival pockets, a gel drug (1.2% concentration of lovastatin) will be applied to the first designated site, and a placebo gel (split-mouth design) will be applied to the second site.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- patients generally healthy, non-smokers, diagnosed with periodontal disease (Experimental): Test side- gingival pocket that meets the inclusion criteria and to which a gel containing 1.2% lovastatin will be assigned in patients generally healthy, non-smokers, diagnosed with periodontitis.
  Interventions: Drug: Subgingival application of 1.2% lovastatin
- Generally healthy patients active smokers with periodontits (Experimental): Test side- gingival pocket that meets the inclusion criteria and to which a gel containing 1.2% lovastatin will be assigned in patients generally healthy,smokers, diagnosed with periodontitis.
  Interventions: Drug: Subgingival application of 1.2% lovastatin
- Generally healthy patients, active smokers with periodontits (Placebo Comparator): control side: gingival pocket that meets the inclusion criteria and to which a placebo gel in patients generally healthy, smokers, diagnosed with periodontitis.
  Interventions: Drug: Subgingival application of placebo gel
- patients generally healthy, non-smokers, diagnosed with periodontitis (Placebo Comparator): control side: gingival pocket that meets the inclusion criteria and to which a placebo gel in patients generally healthy, non-smokers, diagnosed with periodontitis.
  Interventions: Drug: Subgingival application of placebo gel

INTERVENTIONS:
Drug: Subgingival application of 1.2% lovastatin — Each patient will be assigned 2 sites that meet the inclusion criteria. After the SRP (scaling, root planing) procedure is applied within the qualified gingival pockets, a gel drug (1.2% concentration of lovastatin) will be applied to one site selected by randomization.
  Arms: Generally healthy patients active smokers with periodontits; patients generally healthy, non-smokers, diagnosed with periodontal disease
Drug: Subgingival application of placebo gel — Each patient will be assigned 2 sites that meet inclusion criteria. After the SRP procedure (scaling, root planing) procedure is applied within qualified gingival pockets, placebo gel will be applied to one site selected by randomization.
  Arms: Generally healthy patients, active smokers with periodontits; patients generally healthy, non-smokers, diagnosed with periodontitis

SUMMARY:
The aim of the study is to evaluate how a gel (1.2% lovastatin) applied under the gum improves the results of classic periodontal treatment (SRP-scaling, root planing).

The study involves two groups of adults diagnosed with periodontitis: the first group consists of generally healthy individuals who do not smoke tobacco. The second group consists of generally healthy individuals who have been smoking for at least 5 years. Before the study begins, each participant will undergo gum health measurements. Changes in these parameters will be monitored throughout the study. Two teeth will be selected for each participant:

* a gel containing the medication will be applied under the gum of one tooth
* a gel that looks similar to the medication but does not contain any medicinal substance will be applied under the gum of the second tooth.

Before applying the gel, each participant will undergo subgingival cleaning (SRP) to remove any debris that may prevent the medicine from working.

The study will last six months.

Expected results:

* all participants will experience an improvement in the condition of their gums after treatment
* the effect of treatment will be better in non-smokers than in smokers
* the treatment outcome will be better in the area where the medicated gel was applied compared to areas where the gel without medicinal substances was applied.

ELIGIBILITY:
Inclusion Criteria:

* generally healthy patients
* diagnosed periodontal disease (at least one pair of non-adjacent sites with PD≥5 mm or CAL ≥4 mm and vertical bone loss ≥ 3 mm)
* no history of periodontal disease treatment
* no history of antibiotic use in the past 6 months
* an eligible tooth must be alive, with no history of endodontic treatment
* non-smoking (group I) or active smokers (group 2)

Exclusion Criteria:

* Statin allergy
* receiving systemic statin therapy,
* alcoholics
* immunocompromised patients
* pregnant or breastfeeding women.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-07-11 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Clinical Attachment Level | change from baseline to 6 months after intervention
  the distance between the enamel-cement junction (CEJ) and the bottom of the gingival pocket; expressed in mm
Probing Depth | change from baseline to 6 months after intervention
  the distance between the gingival margin and the bottom of the gingival pocket, measured with a calibrated periodontalprobe, expressed in mm
modified Sulcus Bleeding Index | from baseline to six months after intervention
  an index used to determine the severity of inflammation in the periodontal tissues; determines the percentage of the study area that is inflamed
Plaque Index | from baseline to 6 months after intervention
  an index that evaluates the patient'slevel of oral hygiene on a numerical scale of 1-4

SECONDARY OUTCOMES:
Infrabony Defect Depth | from baseline to six months after intervention
  a parameter measured as the distance from the edge of the alveolar crest to the bottom of the bony defect; assessed on conebeam computed tomography (CBCT) scanning

CONTACTS AND LOCATIONS:
Locations (1):
- Pietrzko Dental Clinic, Bielsko-Biala, Silesian Voivodeship, Poland

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan: Study protocol and Statistical Analysis Plan (2025-10-08): https://cdn.clinicaltrials.gov/large-docs/56/NCT07282756/Prot_SAP_000.pdf
  • Statistical Analysis Plan: Results module (2025-11-28): https://cdn.clinicaltrials.gov/large-docs/56/NCT07282756/SAP_001.pdf
  • Informed Consent Form (2025-10-08): https://cdn.clinicaltrials.gov/large-docs/56/NCT07282756/ICF_002.pdf